CLINICAL TRIAL: NCT01411189
Title: Phase III Open-labeled Study of NPO-11 in Patients Undergoing Therapeutic Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPO-11-02/S-02
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Cancer; Colon Nos Polypectomy Tubular Adenoma; Gastric Adenoma
Keywords: therapeutic upper gastrointestinal endoscopy; percutaneous endoscopic gastrostomy; endoscopic mucosal resection; endoscopic submucosal dissection; PEG; EMR; ESD; endoscopic hemostasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Menthol (Other): 20 mL NPO-11
  Interventions: Drug: Menthol

INTERVENTIONS:
Drug: Menthol — 20 mL NPO-11 in prefilled syringe

SUMMARY:
Patients who require therapeutic upper gastrointestinal endoscopy, such as polypectomy, endoscopic hemostasis, percutaneous endoscopic gastrostomy (PEG), endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD), will receive an intragastric spraying of NPO-11. The efficacy of NPO-11 as an anti-peristaltic agent for the endoscopic therapeutic procedures will be evaluated based on the proportion of patients with suppressed gastric peristalsis during the procedures. The degree of gastric peristalsis is assessed by an independent committee.

The safety of NPO-11 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and seven days after administration.

ELIGIBILITY:
Inclusion Criteria:

Inpatients or outpatients of either sex who require therapeutic upper gastrointestinal endoscopy and meet criteria (1), (4), (6) and one from (2), (3) or (5) in the study. Patients have to provide written informed consent for voluntary participation in the study. The criteria (2) to (4) will be confirmed by the endoscopic observation just before starting the intended treatment.

1. Patients who require therapeutic upper gastrointestinal endoscopy (polypectomy, endoscopic hemostasis, PEG, EMR and ESD)
2. Patients with a differentiated-type intramucosal gastric cancer located in the upper or middle third of the stomach (≤2 cm in size, no ulcer finding, EMR or ESD)
3. Patients with a gastric adenoma (≤2 cm in size, no ulcer finding, EMR or ESD)
4. Patients with an a single intended lesion for the treatment
5. Patients without experience of PEG tube placement in case of PEG tube placement
6. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study beforehand. The criteria (3) and (4) will be confirmed by the endoscopic observation just before starting the intended treatment.

1. Patients with a history of surgery to the upper gastrointestinal tract
2. Patients who require emergency endoscopy
3. Patients with severe gastric stenosis or deformation which makes observation of gastric peristalsis difficult
4. Patients who require emergency endoscopic treatment except for the intended lesion
5. Patients with an ongoing cancer treatment (chemotherapy or radiotherapy)
6. Patients with pacemaker
7. Patients with known bleeding tendency or Patients with difficulty of antithrombogenic agents withdrawal
8. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil
9. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
10. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
11. Patients otherwise ineligible for participation in the study in the investigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients had no or mild peristalsis during the therapeutic procedures | 60 minutes
  No or mild gastric peristalsis is defined as when patients have no or suppressed gastric peristalsis during the therapeutic procedure (for 45 s). The degree of gastric peristalsis in the time periods is assessed by an independent committee.

SECONDARY OUTCOMES:
Duration of peristalsis-suppressing effect | 60 minutes
Difficulty level of the therapeutic procedure | 60 minutes
Adverse events and adverse drug reactions | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Tokyo, Japan